CLINICAL TRIAL: NCT03214510
Title: Randomized, Unblinded, Phase III Trial of Thoracic Epidural Analgesia Versus Four-Quadrant Transversus Abdominus Plane Block in Oncologic Open-Incision Liver Surgery
Brief Title: Thoracic Epidural Analgesia or Four-Quadrant Transversus Abdominus Plane Block in Reducing Pain in Patients Undergoing Liver Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-1111; NCI-2018-01124 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1111 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Liver and Intrahepatic Bile Duct Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — Bupivacaine; Fentanyl; Hydromorphone; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (TAE) (Experimental): Patients undergo placement of thoracic epidural catheter before surgery. Patients receive hydromorphone hydrochloride and bupivacaine via thoracic epidural catheter every 10 minutes or 3 hours as needed. Patients may receive fentanyl and bupivacaine or plain bupivacaine via thoracic epidural catheter.
  Interventions: Drug: Bupivacaine; Drug: Fentanyl; Drug: Hydromorphone Hydrochloride; Device: Implanted Medical Device; Behavioral: Questionnaire
- Arm II (TAP) (Experimental): Patients undergo placement of ultrasound-guided, four-quadrant transversus abdominus plane block. Patients receive plain bupivacaine and liposomal bupivacaine via TAP block.
  Interventions: Drug: Bupivacaine; Device: Implanted Medical Device; Drug: Liposomal Bupivacaine; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Bupivacaine — Given via thoracic epidural catheter or TAP block
  Other Names: AH 250
Drug: Fentanyl — Given via thoracic epidural catheter
  Other Names: Abstral; Duragesic
  Arms: Arm I (TAE)
Drug: Hydromorphone Hydrochloride — Given via thoracic epidural catheter
  Other Names: Dilaudid; Dilaudid HP; Dimorphone; Exalgo; Hydromorphone; Hydrostat; Hymorphan; Laudicon; Novolauden
  Arms: Arm I (TAE)
Device: Implanted Medical Device — Undergo placement of thoracic epidural catheter
  Other Names: IMPLANTED
  Arms: Arm I (TAE)
Device: Implanted Medical Device — Undergo placement of ultrasound-guided, four-quadrant transversus abdominus plane block
  Other Names: IMPLANTED
  Arms: Arm II (TAP)
Drug: Liposomal Bupivacaine — Given via TAP block
  Other Names: Bupivacaine Liposome Injectable Suspension; Exparel
  Arms: Arm II (TAP)
Behavioral: Questionnaire — Ancillary studies
  Other Names: Questionnaires

SUMMARY:
This phase III trial studies how well thoracic epidural analgesia or four-quadrant transversus abdominus plane block works in reducing pain in patients undergoing liver surgery. It is not yet known whether thoracic epidural analgesia or four-quadrant transversus abdominus plane block may help people to recover more completely and more quickly after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare length of hospital stay between patients treated with thoracic epidural analgesia (TEA) versus (vs.) pre-incision ultrasound-guided, four-quadrant transversus abdominus plane (TAP) block after open liver resection within an enhanced recovery program.

SECONDARY OBJECTIVES:

I. To compare the area under the curve of early (0-48 hour) post-operative pain scores and number of patients who experience severe postoperative pain between the TEA and TAP groups.

II. To compare anesthetic-related complication rates and need to change modalities between TEA and TAP groups.

III. To compare surgery-related complications (including 30-day readmission and 90-day mortality rates) between TEA and TAP groups.

IV. To compare return to baseline symptom burden, functional and cognitive status between TEA and TAP groups.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients undergo placement of thoracic epidural catheter before surgery. Patients receive hydromorphone hydrochloride and bupivacaine via thoracic epidural catheter every 10 minutes or 3 hours as needed. Patients may receive fentanyl and bupivacaine or plain bupivacaine via thoracic epidural catheter.

ARM II: Patients undergo placement of ultrasound-guided, four-quadrant transversus abdominus plane block. Patients receive plain bupivacaine and liposomal bupivacaine via TAP block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open liver resection without bowel resection/anastomosis for malignancy at MD Anderson Cancer Center
* Patients must sign a study-specific consent form
* Platelets >= 100,000/ml (within 30 days of surgery)
* International normalized ratio (INR) =< 1.5 (within 30 days of surgery)
* Activated partial thromboplastin time (aPTT) =< 40 (within 30 days of surgery)
* Patients must have no fever or evidence of infection or other coexisting medical condition that would preclude epidural placement

Exclusion Criteria:

* Evidence of severe uncontrolled systemic disease or other comorbidity that precludes liver surgery
* History of chronic narcotic use, defined as 30 days or more of preoperative daily narcotic use, measured from the date of surgery
* Anaphylaxis to local anesthetics or narcotics
* Previous or current neurologic disease affecting the lower hemithorax or below
* Major open abdominal/thoracic surgery in the previous 30 days under general anesthesia
* Technical contraindications to epidural placement: previous thoracic spinal surgery or local skin or soft tissue infection at proposed site for epidural insertion
* Use of therapeutic anticoagulation within 5 days of surgery (not including venous thromboembolism prophylaxis)
* Known bleeding diathesis or coagulopathy
* Psychiatric (untreated or poorly controlled schizophrenia, major depression, or bipolar disorder), or communication (language) barrier that would preclude accurate assessment of postoperative pain and/or ability to answer questionnaires (need to be able to read, comprehend, and answer questions)
* Inability to comply with study and/or follow-up procedures
* Patient refusal to participate in randomization
* Pregnant women are excluded from this study; women of childbearing potential (defined as those who have not undergone defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 12 consecutive months) must agree to practice adequate contraception and to refrain from breast-feeding, as specified in the informed consent
* Patients with obvious unresectable disease prior to signing informed consent
* Patients with previous ventral hernia repair, cosmetic abdominoplasty or anterior abdominal wall reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Total length of inpatient stay | Up to 5 years
  Will be recorded and compared between groups. Will be summarized using descriptive statistics including mean, standard deviation, median and range. Will be compared with 2-sample t- tests, Mann Whitney U tests or Wilcoxon rank sum tests as indicated.

SECONDARY OUTCOMES:
Early post-operative pain control | Within 48 hours post surgery
  The area under the curve for each patient will be computed using the trapezoidal method using the pain score by time curve as has been done in prior studies of this type at MD Anderson. Will be compared between groups. In addition, the number of patients experiencing severe pain (>= 7/10) during the inpatient recovery period will be compared between study groups. Will be summarized using descriptive statistics including mean, standard deviation, median and range. Will be compared with 2-sample t- tests, Mann Whitney U tests or Wilcoxon rank sum tests as indicated.
Complication rates secondary to the analgesic regimen | Up to 5 years
  Pain control modality complications will be prospectively recorded including epidural hematoma, epidural catheter migration/malfunction, injection/exit site cellulitis, epidural abscess, cerebrospinal fluid leak, prolonged ileus (defined as inability to tolerate regular diet by post operation day 5), imbalance and gait instability, altered mental status and delirium, and need to change pain control modality due to inadequate pain control. The rate of these complications will be compared between study groups. Will be tabulated with frequency and percentages. Will be compared using chi-square test with Fisher's correction as indicated.
Surgical complication rates | Up to 5 years
  Postoperative surgical complications will be prospectively recorded and graded using the Accordian grading scale. Liver surgery specific complications including bile fistula, bleeding requiring transfusion and liver failure will be recorded. 30-day readmission and 90-day mortality will be recorded. The rates of these complications will be compared between study groups. Will be tabulated with frequency and percentages. Will be compared using chi-square test with Fisher's correction as indicated.
Measures of functional recovery | Up to 5 years
  Quality of recovery will be assessed using the MD Anderson Symptom Inventory for gastrointestinal cancer (MDASI-GI) at regimented intervals including preoperative baseline and postoperative inpatient and outpatient recovery, Return to baseline symptoms including return to baseline life interference summary score at 6 weeks postoperatively, measured using the MDASI-GI, will be compared between groups. Likewise, pre- and post-operative physical and cognitive performance recovery will be compared between groups. Will be summarized using descriptive statistics including mean, standard deviation, median and range. Will be compared with 2-sample t- tests, Mann Whitney U tests or Wilcoxon rank sum tests as indicated.

OTHER OUTCOMES:
Time to readiness for RIOT (return to intended oncologic therapy) | Up to 5 years
  Will be tabulated with frequency and percentages. Will be compared using chi-square test with Fisher's correction as indicated. To assess the relationship between study variables and time to event outcomes (such as RIOT), Kaplan-Meier plots and log-rank tests will be used.
Narcotic utilization | Up to 5 years
  Will be summarized using descriptive statistics including mean, standard deviation, median and range. Will be compared with 2-sample t- tests, Mann Whitney U tests or Wilcoxon rank sum tests as indicated.
Compliance with ordering and delivery of Enhanced Recovery After Surgery program elements | Up to 5 years
  Will be tabulated with frequency and percentages. Will be compared using chi-square test with Fisher's correction as indicated.
Cost of perioperative care | Up to 5 years
  Will be summarized using descriptive statistics including mean, standard deviation, median and range. Will be compared with 2-sample t- tests, Mann Whitney U tests or Wilcoxon rank sum tests as indicated.
Biologic inflammatory markers | Up to 5 years
  Will be summarized using descriptive statistics including mean, standard deviation, median and range. Will be compared with 2-sample t- tests, Mann Whitney U tests or Wilcoxon rank sum tests as indicated.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E. Newhook, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org